CLINICAL TRIAL: NCT06801847
Title: Post-partum Depression in Kentucky: A Community Based Intervention and a Novel AI-powered Screening Tool
Brief Title: Exercise and Socialization in Post-partum Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment
Sponsor: Laura Peterson-Brown (Other)
Responsible Party: Sponsor-Investigator, Laura Peterson-Brown, Post-Doc Scholar, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99825
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Post Partum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Socialization only (Active Comparator)
  Interventions: Behavioral: Socialization
- Socialization and walking (Active Comparator)
  Interventions: Behavioral: Socialization; Behavioral: Walking
- Socialization and moderate exercise (Active Comparator)
  Interventions: Behavioral: Socialization; Behavioral: Moderate Exercise

INTERVENTIONS:
Behavioral: Socialization — Socialization lasting from 30-60 minutes each session
Behavioral: Walking — Twice weekly walking (30 minutes)
  Arms: Socialization and walking
Behavioral: Moderate Exercise — Twice weekly moderate exercise (30 minutes)
  Arms: Socialization and moderate exercise

SUMMARY:
This community-engaged research project aims to address the critical need for alternative treatments of post-partum depression (PPD). The goal of this research is to investigate the efficacy of a novel 8-week intervention combing exercise with social support to reduce PPD symptoms. It is hypothesized that exercise in addition to social support will more effectively reduce PPD symptom severity compared to social support alone. By collaborating with PPD mothers, clinicians, researchers, and local fitness instructors, the researchers aim to develop an intervention that is accessible, culturally appropriate, effective, and increases treatment adherence. Additionally, the researchers will investigate if mother-infant interactions during exercise can enhance bonding, thereby reducing the detrimental effects of maternal PPD on their off-spring.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years old
* Two-weeks to 12 months post-partum
* EPDS over 10
* Read and Speak English
* Willing to supply contact information for their clinician and consent to their clinician being contacted in the event their depression worsens.

Exclusion Criteria:

* Use of anti-depression medication(s) at time of enrollment
* Unable to give consent
* Prisoner, parolee, state probationer, or awaiting sentence for a felony conviction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-28 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in Edinburgh Post-natal Depression Scale (EPDS) score | Baseline, 4 weeks, 8 weeks
  EPDS scores range between 0 and 30.
  EDPS depression ranking system:
  * 0 to 6: No depression or minimal depression
  * 7 to 13: Mild depression
  * 14 to 19: Moderate Depression
  * 20 to 30: Severe Depression

SECONDARY OUTCOMES:
Change in Mother-Infant Bonding Questionnaire (MIBQ) score | Baseline, 4 weeks, 8 weeks
  MIBQ scores are between 0 and 24. Higher score indicates poor mother-baby bonding.

CONTACTS AND LOCATIONS:
Overall Officials: Laura P Brown, PhD, Principal Investigator — University of Kentucky

IPD SHARING:
Plan to Share IPD: No